CLINICAL TRIAL: NCT05637268
Title: Carrelizumab Combined With Chemotherapy for Adjuvant Therapy of Node-positive Thoracic Esophageal Squamous Cell Carcinoma: a One-arm, Phase II Clinical Study
Brief Title: Carrelizumab Combined With Chemotherapy for Adjuvant Therapy of Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Peng Tang, Director, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Peng Tang
Record Dates: First submitted 2022-11-14; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; Long-Term Synaptic Depression; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Treatment with camrelizumab combined with chemotherapy was planned for 4 to 6 cycles, after which carrilizumab monotherapy was maintained until disease progression, unacceptable toxicity, or patient withdrawal.
  A total of 4 to 6 cycles, after carrilizumab maintenance treatment for one year.
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg iv q2w
  Other Names: Suzhou Shengdia Biological Medicine Co., LTD
Drug: Paclitaxel — 150mg/m² iv d1 q2w
Drug: Cisplatin — 50 mg/m² iv d2 q2w

SUMMARY:
This is a single-arm, open, exploratory clinical study to evaluate the efficacy and safety of camrelizumab combined with chemotherapy for adjuvant treatment of nodal positive thoracic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Treatment with carrilizumab combined with chemotherapy was planned for 4 to 6 cycles, after which carrilizumab monotherapy was maintained until disease progression, unacceptable toxicity, or patient withdrawal.

vial card Rayleigh bead sheet resistance: intravenous drip, fixed dose of 200 mg, with 30 minutes to an intravenous drip

(The overall infusion time including the flushing time shall be no less than 20 minutes, no longer than 60 minutes), Day 1, every repeat once every 2 weeks.

paclitaxel: 150 mg/m2, intravenous drip for 30 minutes, 1 day, every 14 days for a cycle.

cisplatin: 50 mg/m2, 2 days, every 14 days for a cycle.

A total of 4 to 6 cycles, after carrilizumab maintenance treatment for one year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed thoracic esophageal squamous cell carcinoma (after R0 resection);
* Lymph node metastases without distant metastases (pM0);
* ECOG PS score: 0 ~ 1
* The enrolled patients were expected to tolerate the combination therapy and survive for more than 6 months.
* The functions of vital organs meet the following requirements (excluding the use of any blood components and cell growth factors within 14 days): - Neutrophils 1.5×10⁹/L - platelet count 100×10⁹ /L - hemoglobin 5.6 mmol/L (9g/dL); Liver and kidney function: - Serum creatinine (SCr) 1.5 times the upper limit of normal (ULN) or creatinine clearance 50 ml/min(Cockcroft-Gault formula); - Upper limit of normal 1.5 times total bilirubin (TBIL) (ULN); - 2.5 times the upper limit of normal (ULN) for aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels; Urine protein <2 +; If the urine protein is ≥2+, the 24-hour urine egg white quantification shows that the protein must be ≤1g
* Coagulation function is normal, no active bleeding and thrombotic disease
* Non-surgical sterilization or female patients of childbearing age who are required to use a medically approved contraceptive method (such as an IUD, birth control pill or condom) during the study treatment period and for 3 months after the study treatment period ends; Female patients of childbearing age who were not surgically sterilized must have a negative serum or urine HCG test within 7 days prior to study enrollment; And it must be non-lactation; Male patients with non-surgical sterilization or of childbearing age need to consent to use a medically approved contraceptive method with their spouse during the study treatment period and for 3 months after the study treatment period ends
* The subjects voluntarily participated in the study with good compliance and safety and survival follow-up

Exclusion Criteria:

* Previous radiotherapy, chemotherapy, concurrent chemoradiotherapy and immunotherapy or other targeted therapy;
* Imaging evidence of distant metastasis;
* Patients with esophageal squamous cell carcinoma after R1 or R2 resection;
* The subject has had or co-had other malignancies (except cured basal cell carcinoma of the skin and cervical carcinoma in situ);
* Patients who had received carrilizumab or other PD-1/PD-L1 treatment in the past could not be enrolled; The subject is known to have a prior allergy to macromolecular protein preparations, or is known to be allergic to any carrilizumab, purple or platinum components;
* Subject has any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with purpura or complete remission of childhood asthma without any intervention as adults could be included; Patients with asthma requiring medical intervention with bronchodilators were not included);
* Subjects who were taking immunosuppressant or systemic or absorbable topical hormone therapy for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormone) and continued to use it within 2 weeks prior to enrollment;
* Ascites or pleural effusion with clinical symptoms, requiring therapeutic puncture or drainage;
* Patients with poorly controlled cardiac clinical symptoms or diseases, such as :(1) heart failure of NYHA2 or above, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
* Abnormal coagulation function (PT>16s APTT>43s TT>21s Fbg>2g/L), bleeding inclination or receiving thrombolytic or anticoagulant therapy;
* Subjects with active infection or unexplained fever >38.5 degrees prior to initial administration during screening (subjects with tumor-related fever, as determined by the investigator, could be enrolled);
* Abdominal fistula and gastrointestinal perforation or abdominal abscess occurred less than 4 weeks before medication;
* Patients with previous or current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia and severe impairment of lung function;
* Subjects with congenital or acquired immune dysfunction, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA 10 /ml; Hepatitis C reference: HCV RNA 10 3 /ml); Chronic hepatitis B virus carriers with HBV DNA<2000 IU/ml(< 104 copies /ml) must also receive antiviral therapy during the trial to be enrolled;
* Subjects are participating in other clinical studies or less than 1 month after the end of the previous clinical study; Subjects may receive other systemic antitumor therapies during the study;
* Live vaccine was administered less than 4 weeks before or possibly during the study period;
* The subject has a known history of psychotropic substance abuse, alcohol abuse or drug use;
* The researcher considers that the subjects should be excluded from the study. For example, the researcher judges that the subjects have other factors that may cause the study to be terminated, such as other serious diseases (including mental illness). Concomitant treatment is required, there are serious laboratory abnormalities associated with family or social factors that may affect the safety of the subject or the collection of data and samples.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | 8 weeks
  The probability of 3-year disease-free survival

SECONDARY OUTCOMES:
DFS | From date of randomization until the date of first documented progression, assessed up to 60 months
  disease-free survival
3 years OS rate | 8 weeks
  The probability of 3-year overall survival
5 years OS rate | 8 weeks
  The probability of 5-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Peng Tang, archiater, Study Chair — Affiliated Cancer Hospital of Tianjin Medical University
Locations (1):
- Affiliated Cancer Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No